CLINICAL TRIAL: NCT02896920
Title: Canadian Humira Post Marketing Observational Epidemiological Study : Assessing Humira Real-life Effectiveness and Impact on Hidradenitis Suppurativa (HS) Burden of Illness and Health Care Resources Utilization
Brief Title: Canadian Humira Post Marketing Observational Epidemiological Study : Assessing Humira Real-life Effectiveness and Impact on HS Burden of Illness
Acronym: SOLACE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-696
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Hidradenitis Suppurativa (HS); Humira®; Canada
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants receiving adalimumab/ Humira®: Participants with HS for whom a change in treatment to Humira® is made by the treating physician

SUMMARY:
This study assesses Humira's® real-life effectiveness in the management of dermatological manifestations of moderate to severe Hidradenitis Suppurativa (HS).

ELIGIBILITY:
Inclusion Criteria:

* Has a clinical diagnosis of moderate to severe HS according to the treating physician judgment
* Need a change in ongoing therapy for any reason, but not limited to inadequate response, intolerance, sub-optimal compliance, or patient preference. Patient will be approached to participate in the study after a decision to change patient's therapy for Humira® is made by the treating physician.
* Has provided written informed consent (Patient Authorization) for participation in the study

Exclusion Criteria:

* Is participating in a clinical interventional study
* Was treated with Humira®, or any other biologic agents for HS prior to baseline visit
* Has any other active skin disease or condition that, in the opinion of the treating physician, prohibits the patient from participating in the study or obscures the assessment of the treatment of HS

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with moderate or severe HS
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving clinical response using the Hidradenitis Suppurativa Clinical Response measure (HiSCR) at week 24 | At Week 24
  The HiSCR measure is defined as at least a 50% reduction in the Abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count relative to baseline.

SECONDARY OUTCOMES:
Proportion of participants who experience flare | Up to Week 52
  It is defined as at least 25% increase in AN counts with a minimum increase of 2 relative to baseline
Change from Baseline in Hospital Anxiety and Depression Scale (HADS) | From Week 0 (baseline) to Week 52
  The HADS questionnaire includes 14 questions that evaluate the level of anxiety and depression an HS patient may experience associated with HS. A lower score indicates less severity.
Change from Baseline in International Index of Erectile Function (IIEF) | From Week 0 (baseline) to Week 52
  The IIEF contains 15 questions that were assigned in 5 domains of male sexuality: erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction.
Change from Baseline in Health Care Resource Utilization (HCRU) associated with HS | From Week 0 (baseline) to Week 52
  This will be assessed using a descriptive questionnaire that aimed at measuring the patient's health care resource utilization and economic impact of HS.
Change from Baseline in Patient Global Assessment of HS (HS-PtGA) | From Week 0 (baseline) to Week 52
  The HSPtGA consists in one question that evaluates how one patient ranked the severity of HS at the time of the routine visit.
Proportion of participants achieving clinical response using the Hidradenitis Suppurativa Clinical Response measure (HiSCR) at week 52 | At Week 52
  The HiSCR measure is defined as at least a 50% reduction in the Abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count relative to baseline.
Change from Baseline in Health Utility Index Mark 3 (HUI3) | From Week 0 (baseline) to Week 52
  This is a comprehensive system for measuring health status and health-related quality of life and for producing utility scores.
Change from Baseline in Female Sexual Function Index (FSFI) | From Week 0 (baseline) to Week 52
  The FSFI questionnaire contains 19 questions that describe the female sexual function in 6 domains. The domains are: desire, arousal, lubrication, orgasm, satisfaction, and pain, which can both be evaluated individually and in their entirety.
Proportion of participants who experience worsening of HS by >= 1 Hurley Stage in >= 1 affected anatomic region | Up to Week 52
  This will be done by evaluating the Hurley Stage using the following description:
  Stage I: Abscess formation, single or multiple, without sinus tracts and cicatrization (scarring).
  Stage II: One or more widely separated recurrent abscesses with tract formation and cicatrization (scars).
  Stage III: Multiple interconnected tracts and abscesses across the entire area, with diffuse or near diffuse involvement.
Change from Baseline in Hidradenitis Suppurativa Symptom Assessment (HSSA) | From Week 0 (baseline) to Week 52
  The HSSA questionnaire includes 9 questions that evaluate the symptoms an HS participant may experience associated with HS.
Change from Baseline in Hidradenitis Suppurativa Impact Assessment (HSIA) | From Week 0 (baseline) to Week 52
  The HSIA questionnaire includes 18 questions that evaluate the impacts an HS participant may experience associated with HS.
Change from Baseline in Work Productivity and Activity Impairment Questionnaire: Specific Health Problem V2.0 (WPAI: SHP) | From Week 0 (baseline) to Week 52
  The WPAI: SHP evaluates four areas: percent work time missed due to HS, percent impairment while working due to HS, percent overall work impairment due to HS, and percent activity impairment due to HS.
Number of days where participants experience HS flare-up | Up to Week 52
  It is calculated from the day when flare is observed to the day prior to the observation that flare is no longer present. Of note, there could be multiple periods that flares are observed, in which case, the total days from the multiple periods will be used.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (22):
- Canada (22):
  - Institute for Skin Advancement /ID# 152448, Calgary, Alberta
  - Alberta DermaSurgery Centre /ID# 153834, Edmonton, Alberta
  - Jason Ronald Sneath Medical Co /ID# 152462, Brandon, Manitoba
  - Winnipeg Clinic, Manitoba, CA /ID# 153830, Winnipeg, Manitoba
  - Wiseman Dermatology Research /ID# 153835, Winnipeg, Manitoba
  - Dr. Irina Turchin PC Inc. /ID# 152464, Fredericton, New Brunswick
  - Karma Clinical Trials /ID# 152444, St. John's, Newfoundland and Labrador
  - NewLab Clinical Research Inc. /ID# 152438, St. John's, Newfoundland and Labrador
  - Dr. Brown-Maher PMC INC. /ID# 152407, St. John's, Newfoundland and Labrador
  - Eastern Canada Cutaneous Resea /ID# 153832, Halifax, Nova Scotia
  - SimcoMed Health Ltd /ID# 152445, Barrie, Ontario
  - Dr. Wei Jing Loo Medicine Prof /ID# 157923, London, Ontario
  - Lynderm Research Inc. /ID# 152436, Markham, Ontario
  - SKIN Centre for Dermatology /ID# 152457, Peterborough, Ontario
  - York Dermatology Center /ID# 152403, Richmond Hill, Ontario
  - Niakosari Medicine Professional Corporation /ID# 157851, Toronto, Ontario
  - K. Papp Clinical Research /ID# 152446, Waterloo, Ontario
  - Dr. Isabelle Delorme Inc. /ID# 152408, Drummondville, Quebec
  - Clinique D /ID# 152406, Laval, Quebec
  - Dre. Angelique Gagne-Henley /ID# 152611, Saint-Jérôme, Quebec
  - Dermatologie Sima Inc. /ID# 152443, Verdun, Quebec
  - Hopital St-Sacrement /ID# 152456, Québec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P15-696.pdf